CLINICAL TRIAL: NCT03694171
Title: Access to Care and Prognosis in Elderly Cancer Patients: Analysis of Determinants Using Data From Cancer Registries and Cohort Studies in Gironde, French Department
Brief Title: Access to Care and Prognosis in Elderly With Cancer (INCAPAC Study)
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University of Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: IB2013 INCAPAC
Record Dates: First submitted 2018-09-21; First posted 2018-10-03 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Cancer
Keywords: Elderly; Cancer; Cohort study; Cancer registry; Access to care; Cancer stage; Cancer treatment; Prognosis; Functional decline; Survival
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Older patients with cancer: Subjects i) aged 65 years and over from the PAQUID, the 3City or the AMI study; ii) alive on January 1st 2005 (common start date of tumor recording); iii) resident in Gironde; and iv) with a validated cancer diagnosis recorded in one of the cancer registries from January 1st 2005 to December 31st 2014. We included all invasive malignant tumors (including skin tumors) and benign tumors of the central nervous system. For patients with multiple tumors, only one was considered: i) the first one diagnosed if there were several tumors with a minimum of a 6 months interval between their diagnosis, ii) the one with the worse prognosis if there were several tumors diagnosed within less than 6 months.
  Interventions: Other: Any cancer treatment

INTERVENTIONS:
Other: Any cancer treatment

SUMMARY:
The growing incidence of cancer associated to an aging population represents an epidemiologic reality that requires questioning access to care and prognosis in elderly with cancer, for which disparities have been highlighted. However, generally speaking, studies are limited in that they overlook geriatric-specific factors. The aim of this work was to study sociodemographic, socioeconomic and clinical determinants of access to care (cancer stage, cancer treatment) and prognosis (functional decline, survival) in elderly cancer patients.

DETAILED DESCRIPTION:
The French department of Gironde (1.5 million inhabitants) is covered by cancer registries. In addition, three cohorts were initiated in Gironde on cerebral and functional aging that enrolled subjects aged 65 years and over: the PAQUID study (1988), the 3-City study (1999), and the AMI study (2007). In these cohorts, a large amount of individual data on the participants has been collected longitudinally at different follow-up visits, conducted every two or three years.

Using cancer registries, older subjects with cancer were identified in the cohort studies. Subjects were included if they presented the following: i) aged 65 years and over from one of the three cohorts, ii) alive on January 1st 2005 (common start date for tumor recording) and resident in Gironde, and iii) with a validated cancer diagnosis recorded in one of the cancer registries from January 1st 2005 to December 31st 2014. All tumors for which data is annually sent by cancer registries to the International Agency for Research of Cancer were included: invasive malignant tumors and benign tumors of the central nervous system. As the incidence of skin tumors in older cancer patients is high, they were also included. For patients with multiple tumors, only one was considered: either the first one diagnosed if there were several tumors with a minimum of a 6 months interval between their diagnosis, or the one with the worse prognosis if there were several tumors diagnosed within 6 months.

In order to not consider information concerning patients' characteristics that was too old, subjects with a delay between the last completed cohort follow-up visit before the cancer diagnosis and the diagnosis of cancer equal or superior to 6 years were excluded.

Variables were extracted from cohorts and registries at different times: cohort inclusion, pre-diagnosis visit, cancer diagnosis or registries follow-up.

ELIGIBILITY:
* Age ≥ 65 years
* Alive on January 1st 2005 ( PAQUID or 3-City cohorts) or included in the AMI cohort study
* Cancer diagnosis recorded in one of the cancer registries in Gironde, French department

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Subjects aged 65 and over with a diagnosis of cancer recorded in one of the cancer registries in Gironde, French department.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simone Mathoulin-Pelissier, MD-PhD, Study Chair — Institut Bergonié
Locations (1):
- Institut Bergonié, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Galvin A, Helmer C, Coureau G, Amadeo B, Joly P, Sabathe C, Monnereau A, Baldi I, Rainfray M, Soubeyran P, Delva F, Mathoulin-Pelissier S. Determinants of cancer treatment and mortality in older cancer patients using a multi-state model: Results from a population-based study (the INCAPAC study). Cancer Epidemiol. 2018 Aug;55:39-44. doi: 10.1016/j.canep.2018.04.013. Epub 2018 May 25. PMID 29763754
- [Result] Galvin A, Delva F, Helmer C, Rainfray M, Bellera C, Rondeau V, Soubeyran P, Coureau G, Mathoulin-Pelissier S. Sociodemographic, socioeconomic, and clinical determinants of survival in patients with cancer: A systematic review of the literature focused on the elderly. J Geriatr Oncol. 2018 Jan;9(1):6-14. doi: 10.1016/j.jgo.2017.07.007. Epub 2017 Oct 10. PMID 29030150

RESULTS

PARTICIPANT FLOW:
Groups:
- Older Patients With Cancer: Subjects i) aged 65 years and over from the PAQUID, the 3City or the AMI study; ii) alive on January 1st 2005 (common start date of tumor recording); iii) resident in Gironde; and iv) with a validated cancer diagnosis recorded in one of the cancer registries from January 1st 2005 to December 31st 2014. We included all invasive malignant tumors (including skin tumors) and benign tumors of the central nervous system. For patients with multiple tumors, only one was considered: i) the first one diagnosed if there were several tumors with a minimum of a 6 months interval between their diagnosis, ii) the one with the worse prognosis if there were several tumors diagnosed within less than 6 months.
  Any cancer treatment
Period: Overall Study
Arm/Group | Older Patients With Cancer
Started | 450
Completed | 450
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Older Patients With Cancer
Number analyzed (Participants) | 450
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 450
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204
  Male | 246
Region of Enrollment [Number; unit: participants]
  France | 450

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Being Receiving Treatment Administration After Diagnosis
Description: Treatment administration was defined as any cancer treatment (versus no treatment) including curative, palliative and symptomatic treatments.
  This information was registered by registries and qualified as unknown when no information was available about treatment receipt.
Time Frame: At diagnosis
Measure: Count of Participants; unit: Participants
Arm/Group | Older Patients With Cancer
Number analyzed (Participants) | 450
Participants | 372

2. Primary Outcome: The Probability of Being Dead at One Year
Description: The probability of being dead with or without receiving cancer treatment at least once (death)
Time Frame: one year after diagnosis
Measure: Number; unit: percentage of participants
Arm/Group | Older Patients With Cancer
Number analyzed (Participants) | 450
percentage of participants | 35.5

ADVERSE EVENTS:
Time Frame: One year Serious and Other (Not Including Serious) Adverse Events were not monitored/assessed
Description: Serious and Other (Not Including Serious) Adverse Events were not monitored/assessed
Arm/Group | Older Patients With Cancer
All-Cause Mortality (participants affected / at risk) | 160/450
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes